CLINICAL TRIAL: NCT04070339
Title: A Study on Cerebral Blood Flow Velocity Reference Values Considering Age, Blood Pressure and Carbon Dioxide Partial Pressure i n Small Children: a Prospective Observational Study
Brief Title: Cerebral Blood Flow Using Transfontanelle Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Other Study IDs: 1908-111-105
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Blood Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transfontanelle ultrasound — cerebral blood flow investigation using transfontanelle ultrasound

SUMMARY:
We planned to evaluate cerebral blood flow and its association with age, blood pressure, and end tidal carbon dioxide in small pediatric using transfontanelle ultrasound during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia

Exclusion Criteria:

* patients with hydrocephalus, brain tumor

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatrics including preterm neonates undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
cerebral blood flow | from anesthetic induction to postanesthesia care unit discharge, an average of 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided